CLINICAL TRIAL: NCT05940168
Title: Feasibility, Effectiveness and Qualitative Experiences of Internet-delivered ACT for Parents of Children With Disabilities
Brief Title: Internet-delivered ACT (I-Navigator ACT) for Parents of Children With Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Forte (Industry); Stiftelsen Frimurarna Barnhuset (Unknown)
Responsible Party: Principal Investigator, Tatja Hirvikoski, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I-Navigator ACT
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Parents; Stress, Psychological; Anxiety; Depression; Neurodevelopmental Disorders; Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Intellectual Disability; Physical Disability; Traumatic Brain Injury
Keywords: Acceptance and Commitment Therapy; Mindfulness; Experiential avoidance; Autistic children; Parental stress; Disability; Mental health; Telehealth; Internet delivered treatment; Randomized controlled trial; Group therapy; Families; Qualitative study; Interviews
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Depression; Neurodevelopmental Disorders; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Intellectual Disability; Brain Injuries, Traumatic; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The main study in this project (Study 2) is a randomized controlled trial in which the participants are randomly assigned either a group intervention (Navigator ACT), or an internet-delivered ACT intervention (I-Navigator ACT). No treatment-as-usual (TAU) or wait-list control groups are included in this model.
Who Masked: Participant, Care Provider
Masking Description: Masking at baseline for both participant and care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigator ACT group (Active Comparator): This is a manualized Acceptance and Commitment Therapy group-intervention for 8-16 parents of children with disabilities. The intervention consists of five group sessions with different themes, as well as a booster-session at three months after the fifth session. The intervention is held by two group leaders.
  Interventions: Behavioral: Navigator ACT group
- I-Navigator ACT (Experimental): This intervention is an internet-delivered version of the manualized Acceptance and Commitment Therapy group. The internet-delivered version is given as an individual treatment via a secure online treatment platform. It consists of ten separate chapters or modules. The duration of the intervention is 10-12 weeks, with a individual follow up-session by phone or video at three months after completion.
  Interventions: Behavioral: I-Navigator ACT

INTERVENTIONS:
Behavioral: I-Navigator ACT — The intervention is an internet-delivered ten module Acceptance and Commitment Therapy treatment program for stressed and distressed parents of children with disabilities. The contents of the program is mostly text based, but also includes videos, mindfulness exercises and written exercises, as well as homework between modules.
  Arms: I-Navigator ACT
Behavioral: Navigator ACT group — The intervention is a five session Acceptance and Commitment Therapy group treatment for stressed and distressed parents of children with disabilities. All five sessions have different themes and are held by two group leaders. Sessions are around two and a half hours long. Homework is given between sessions.
  Arms: Navigator ACT group

SUMMARY:
The purpose of the project is to evaluate the feasibility, acceptability, and effectiveness of the internet-delivered Acceptance and Commitment Therapy treatment (I-Navigator ACT) for parents who experience stress, distress, depression or anxiety that may be associated with being a parent of a child with disabilities. The project consists of three studies:

Study 1: An open feasibility trial in which parents participate in an individual, clinician-supported internet-delivered Acceptance and Commitment Therapy treatment.

Study 2: A randomized controlled trial in which participants are randomly assigned either:

1. Navigator ACT group treatment, where parents participate in an Acceptance and Commitment Therapy group together with other parents, led by two group leaders, or
2. I-Navigator ACT internet-delivered Acceptance and Commitment Therapy treatment, where the parent participates on their own, coached by a clinician via a message function.

Study 3: A qualitative study in which a smaller sample of parents from the open feasibility trial participate in semi-structured interviews. The interviews take place after the parents have completed I-Navigator ACT.

All three studies are conducted in a clinical health care context.

DETAILED DESCRIPTION:
Internet Navigator ACT (I-Navigator ACT) is an individual, internet-delivered Acceptance and Commitment Therapy (ACT) treatment, adapted from the manualized ACT group Navigator ACT for parents of children with disabilities. The purpose of I-Navigator ACT is to provide a treatment option that isn't bound by geography, especially beneficial for patients who have limited access to in-person support and care. I-Navigator ACT was developed with a co-creation approach, which included pilot testing with a small group of parents to gather their detailed feedback. Their feedback was considered for refining the treatment.

I-Navigator ACT consists of ten online modules with different themes based on ACT processes. Participants receive weekly written support from an experienced clinician (coach), via a message function. The program is available through the Swedish national platform for internet-delivered treatments (1177.se).

There are three studies planned in this project. The first study (Study 1) will be conducted as a open feasibility trial, in which all participating parents after enrolment and inclusion (via telephone or video call) will be allocated to the I-Navigator ACT treatment. The main purpose of this study is to evaluate feasibility and acceptability of the treatment. Feasibility is measured through treatment completion, treatment credibility and expectation, as well as treatment satisfaction. Preliminary outcomes regarding effectiveness will also be evaluated in this study. Participants are being assessed at pre-treatment, post-treatment, and three months post-treatment.

The second study (Study 2) will be conducted as a randomized controlled trial with two treatment arms. The randomized controlled trial is conducted to evaluate the effectiveness of the I-Navigator ACT treatment compared to the Navigator ACT group treatment. After enrolment and screening via telephone or video call, eligible participants are invited to an information meeting. Once the participants have given their informed consent and completed pre-treatment assessments, they are randomly assigned either the five-session Navigator ACT group, or the I-Navigator ACT treatment. The treatments run parallel during the same semester, and participants are being assessed at the same time points (pre-treatment, post-treatment, and three months post treatment). Effectiveness will be evaluated through the primary outcome measure of acceptance and action-based skills, and secondary outcome measures parental stress, depression and anxiety symptoms, experiential avoidance, mindfulness-based skills, and parent-rated child behavioral problems.

The third and final study (Study 3) will be a qualitative study based on semi-structured interviews, and will be utilizing a thematic content analysis. The interviews will mainly focus on the experience of participating in an internet-delivered ACT treatment for parents.

Data collection commenced in early spring of 2021 (beginning with the open feasibility study) and is projected to be completed by November 2023. N = 32 participants have been allocated to treatment in the open feasibility study, whereas n = 134 participants have been allocated to treatment in the RCT. Nine parents have participated in qualitative interviews.

ELIGIBILITY:
Inclusion Criteria (in all studies):

* Being a parent of at least one child (4-17 years of age) with any or several of the following disabilities: autism spectrum disorder, attention deficit hyperactivity disorder, intellectual disability, physical disability (eg cerebral palsy), traumatic brain injury and/or a profund and multiple intellectual disability (PMID)
* Experiencing stress, distress, depression and/or anxiety that to some extent may be associated with being a parent of a child with a disability
* Having access to a personal computer or tablet with a stable internet connection
* In Study 2 (RCT) also: being able to participate in the group treatment OR the internet-delivered treatment

Exclusion Criteria:

* Currently experiencing a serious mental disorder (eg ongoing psychosis, acute suicidal behaviours) or currently being treated at an in-patient mental health facility
* Not experiencing stress, distress, depression and/or anxiety that to some extent may be associated with being a parent of a child with a disability
* Not being able to read, write or speak the Swedish language
* Not being able to participate in all planned sessions
* Not having access to a personal computer or tablet with a stable internet connection
* In Study 2 (RCT) also: not being able to participate in the group treatment OR the internet-delivered treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Study 1: Treatment completion rate | Participants are assessed during the 10-12 weeks long treatment.
  In this feasibility study (study 1), treatment completion is defined as completing 7 out of 10 intervention sessions/modules. The benchmark for good feasibility is 75% of participants completing the treatment.
Study 2: Changes in parental psychological flexibility and experiential acceptance | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  Parental Acceptance and Action Questionnaire (PAAQ), a scale that targets psychological flexibility and experiential acceptance in the parenting context, i.e., measures to which extent parents' accept inner experiences related to parenting and the readiness to take appropriate and needed action in parenting (commitment to values-based actions). This was originally a 19-item scale.
Study 3: Experiences of participating in an internet-delivered ACT treatment for parents | The interviews are conducted after (circa 3 months) parents have participated in the I-Navigator ACT treatment.
  The semi-structured interviews with parents after they have participated in the I-Navigator ACT treatment are based on the following seven interview questions:
  1. How was your experience participating in I-Navigator ACT?
  2. What aspects of the treatment did you appreciate?
  3. What aspects of the treatment did you appreciate less?
  4. Have you noticed any changes in your life, or everyday life after going through the treatment? Could you describe them?
  5. What aspects of the treatment do you think will be useful to you?
  6. What would you like to change about the treatment?
  7. If you were given the possibility to participate in the treatment but in a different format, eg in a group context, or one-on-one with your care provider in a physical room, what do you think would have been different, and what would be quite similar to your experience? How do you think you would find that?

SECONDARY OUTCOMES:
Study 1: Changes in general stress and parental stress | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  Participants levels of stress and distress are assessed through the Parental Stress Scale (PSS), which is a 18-item psychometric scale (scored 1-5, where 1 indicates that the participant "Completely disagrees" with the statement and 5 indicates that the participant "Completely agrees" with the statement). Low scores indicate low levels of parental stress, whereas high scores indicate high levels of parental stress.
  Another measure of stress is the Perceived Stress Scale 4 Items (PSS-4), which is a 4-item psychometric scale (scored 0-4, where 0 indicates "Never" and 4 indicates "Very often"). Low scores indicate low levels of stress, whereas high scores indicate high levels of stress.
  The PSS measurement scale targets the specific kind of stress experienced by many parents, especially the stress experienced by parents of children with psychological/behavioral problems and children with disabilities. The PSS-4 measurement scale is designed to measure common stress symptoms.
Study 1: Changes in depression and anxiety symptoms | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 items (scored 0-4, where 0 - "Often", and 4 - "Never"), subsequently summarized for an overall score. Low scores indicate none or very mild depressive and/or anxiety symptoms, whereas high scores indicate clinical levels of severe depression and or/anxiety.
Study 1: Changes in mindfulness-based skills | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The Mindfulness Awareness Attention Scale (MAAS), a 15-item scale (scored 1-6, where 1 indicates "Almost always" and 7 indicates "Never") assessing dispositional mindfulness in regards to cognitive, emotional, physical, interpersonal and general domains.
Study 1: Changes in psychological flexibility and experiential acceptance | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The AAQ assessment is intended to measure psychological flexibility and experiential acceptance in a general context. It intends to measure to which extent one accepts inner experiences, and the readiness to take appropriate and needed action in one's life (commitment to values-based actions). AAQ is a 7-item psychometric scale (scored 1-7, where 1 indicates "Never true" and 7 indicates "Always true").
Study 1: Change in child's difficulties and the impact of these difficulties on the child's family | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The Strengths and Difficulties Questionnaire (P4-17 SDQ), a caregiver administered, 25-item extended version of SDQ used for behavior screening of children and adolescents in ages 4-17 years. The SDQ P4-17 covers common areas of emotional and behavioral difficulties and strengths. It also includes a caregiver reported impact and burden assessment.
Study 2: Changes in general stress and parental stress | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  Participants levels of stress and distress are assessed through the Parental Stress Scale (PSS), which is a 18-item psychometric scale (scored 1-5, where 1 indicates that the participant "Completely disagrees" with the statement and 5 indicates that the participant "Completely agrees" with the statement). Low scores indicate low levels of parental stress, whereas high scores indicate high levels of parental stress.
  Another measure of stress is the Perceived Stress Scale 4 Items (PSS-4), which is a 4-item psychometric scale (scored 0-4, where 0 indicates "Never" and 4 indicates "Very often"). Low scores indicate low levels of stress, whereas high scores indicate high levels of stress.
  The PSS measurement scale targets the specific kind of stress experienced by many parents, especially the stress experienced by parents of children with psychological/behavioral problems and children with disabilities. The PSS-4 measurement scale is designed to measure common stress symptoms.
Study 2: Changes in depression and anxiety symptoms | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 items (scored 0-4, where 0 - "Often", and 4 - "Never"), subsequently summarized for an overall score. Low scores indicate none or very mild depressive and/or anxiety symptoms, whereas high scores indicate clinical levels of severe depression and or/anxiety.
Study 2: Changes in mindfulness-based skills | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The Mindfulness Awareness Attention Scale (MAAS), a 15-item scale (scored 1-6, where 1 indicates "Almost always" and 7 indicates "Never") assessing dispositional mindfulness in regards to cognitive, emotional, physical, interpersonal and general domains.
Study 2: Changes in psychological flexibility and experiential acceptance | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The AAQ assessment is intended to measure psychological flexibility and experiential acceptance in a general context. It intends to measure to which extent one accepts inner experiences, and the readiness to take appropriate and needed action in one's life (commitment to values-based actions). AAQ is a 7-item psychometric scale (scored 1-7, where 1 indicates "Never true" and 7 indicates "Always true").
Study 2: Change in child's difficulties and the impact of these difficulties on the child's family | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  The Strengths and Difficulties Questionnaire (P4-17 SDQ), a caregiver administered, 25-item extended version of SDQ used for behavior screening of children and adolescents in ages 4-17 years. The SDQ P4-17 covers common areas of emotional and behavioral difficulties and strengths. It also includes a caregiver reported impact and burden assessment.

OTHER OUTCOMES:
Study 1: Treatment Credibility Scale (TCS) | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), and post-treatment, at the time of completing the intervention (T2).
  As a measure of feasibility, TCS is used to measure the expectation of improvement and treatment credibility. The TCS is a visual analogue scale rated from "Low credibility"/ "Not at all" (0) to "High credibility"/"Very much" (10) and the score calculated is a mean of all items. The TCS was administered after providing thorough information and presentation of the treatment content at baseline and after completion of the treatment. The item wording after adjustment to the current study were: (1) How logical does the treatment seem to you? (2) How confident are you that this treatment will reduce your distress? (3) Would you recommend the treatment to a friend experiencing the same type of distress? (4) How successful do you feel this type of treatment is in improving your psychological health? 5) At this very moment, to what degree has the treatment improved your psychological health?
Study 1: Current Life Situation Form (CLS) | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  Participants complete the Current Life Situation Form in order to collect relevant demographic data, as well as measures on their quality of life. A complete version of the form is administered at the time of inclusion (T1), whereas a shorter version of the form (sans demographic data) is administrered at follow up (T2), (T3).
Study 1: Module Evaluation Form | Participants rate each of every ten modules after each module is completed during the 10-12 weeks of ongoing treatment.
  An 8-item form, scored 1-5 where participants rate the current module.
Study 2: Treatment Credibility Scale (TCS) | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), and post-treatment, at the time of completing the intervention (T2).
  As a measure of feasibility, TCS is used to measure the expectation of improvement and treatment credibility. The TCS is a visual analogue scale rated from "Low credibility"/ "Not at all" (0) to "High credibility"/"Very much" (10) and the score calculated is a mean of all items. The TCS was administered after providing thorough information and presentation of the treatment content at baseline and after completion of the treatment. The item wording after adjustment to the current study were: (1) How logical does the treatment seem to you? (2) How confident are you that this treatment will reduce your distress? (3) Would you recommend the treatment to a friend experiencing the same type of distress? (4) How successful do you feel this type of treatment is in improving your psychological health? 5) At this very moment, to what degree has the treatment improved your psychological health?
Study 2: Current Life Situation Form (CLS) | Participants are assessed at the time of inclusion, circa two weeks prior to the beginning of the intervention (T1), post-treatment, at the time of completing the intervention (T2), and at around three months after completing the intervention (T3)
  Participants complete the Current Life Situation Form in order to collect relevant demographic data, as well as measures on their quality of life. A complete version of the form is administered at the time of inclusion (T1), whereas a shorter version of the form (sans demographic data) is administrered at follow up (T2), (T3).
Study 2: Module Evaluation Form | Participants rate each of every ten modules after each module is completed during the 10-12 weeks of ongoing treatment.
  An 8-item form, scored 1-5 where participants rate the current module.
Study 2 (only): Session Evaluation Form | Participants rate each of every five group sessions after each session is completed during the 10-12 weeks of ongoing treatment.
  An 8-item form, scored 1-5 where participants rate the current group session.

CONTACTS AND LOCATIONS:
Overall Officials: Tatja Hirvikoski, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Habilitering & Hälsa, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No